CLINICAL TRIAL: NCT05427357
Title: Evaluation of The Results of Closed Kinetic Chain Exercises Applied in The Conservative Treatment of Patellofemoral Pain Syndrome by Means of Shear Wave Elastography: A Randomized Controlled Trial
Brief Title: Evaluation of the Results of Closed Kinetic Chain Exercises in Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taksim Egitim ve Arastirma Hastanesi (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Taksim eğitim
Record Dates: First submitted 2022-06-07; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Exercise Training
Keywords: Elastography; exercises; non-selective; pain; patellofemoral
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diseased side of the patellofemoral pain syndrome (PFPS) group (40 knees) (Experimental): Non-selective close kinetic chain exercises and selective close kinetic chain exercises were applied for 6 weeks in diseased side of the PFPS group. Thigh circumference measurement was performed 5-10 cm above the upper pole of the patella. In addition, evaluation was made with visual analog score (VAS) and Lysholm Knee score (LKS). Vastus medialis obliquus (VMO) and vastus lateralis (VL) muscles of the participants were measured with Shear Wave Elastography 1 day before the therapy and 6 weeks after therapy in hospital.
  Interventions: Other: Non-selective closed kinetic chain exercises (NSKCE) and selective closed kinetic chain exercises (SCKCE)
- Healthy side of the patellofemoral pain syndrome (PFPS) group (40 knees) (Experimental): Non-selective close kinetic chain exercises and selective close kinetic chain exercises were applied for 6 weeks in healthy side of the PFPS group. Thigh circumference measurement was performed 5-10 cm above the upper pole of the patella. In addition, evaluation was made with visual analog score (VAS) and Lysholm Knee score (LKS). Vastus medialis obliquus (VMO) and vastus lateralis (VL) muscles of the participants were measured with Shear Wave Elastography 1 day before the therapy and 6 weeks after therapy in hospital.
  Interventions: Other: Non-selective closed kinetic chain exercises (NSKCE) and selective closed kinetic chain exercises (SCKCE)
- Both side of the healthy control group (80 knees) (Other): Non-selective close kinetic chain exercises and selective close kinetic chain exercises were applied for 6 weeks in side of the both side of the healthy control group. Thigh circumference measurement was performed 5-10 cm above the upper pole of the patella. In addition, evaluation was made with visual analog score (VAS) and Lysholm Knee score (LKS). Vastus medialis obliquus (VMO) and vastus lateralis (VL) muscles of the participants were measured with Shear Wave Elastography 1 day before the therapy and 6 weeks after therapy in hospital.
  Interventions: Other: Non-selective closed kinetic chain exercises (NSKCE) and selective closed kinetic chain exercises (SCKCE)

INTERVENTIONS:
Other: Non-selective closed kinetic chain exercises (NSKCE) and selective closed kinetic chain exercises (SCKCE) — Non-selective closed kinetic chain double-leg semi-squat exercise In this exercise, the standing patient leans his or her back against the wall and slides down the wall until the knees are about 45 degrees flexed. Daily program was determined as 5 sessions and 10 repeats. The knee stayed at flexion position for 10 seconds in each repeat, which aimed the contraction of quadriceps muscle. There is a relaxation period for 5 seconds between each repeat.
  Selective closed kinetic chain double-leg semi-squat exercise with hip adduction In this exercise, the standing patient leans his or her back against the wall, forces the knees for adduction by squeezing the pillow placed between the knees and slides down the wall until the knees are about 45 degrees flexed. Daily program was determined as 5 sessions and 10 repeats.

SUMMARY:
Non-selective closed kinetic chain exercises and or selective closed kinetic chain exercises has been shown to increase Vastus medialis obliquus muscle power in patellofemoral pain syndrome. However, the superiority of the exercises to each other has not been shown.

This study aimed to evaluating the effects of different exercises on the stiffness of the Vastus medialis obliquus and vastus lateralis muscles, pain management, functional scores, and thigh circumferences.

DETAILED DESCRIPTION:
This randomized-controlled clinical trial included 40 patients (20 male and 20 female) who were admitted to hospital and who were clinically diagnosed with single-sided patellofemoral pain syndrome (PFPS) and 40 healthy controls (20 male and 20 female). Each group were randomized into subgroups according to diseased side of the PFPS group (40 knees), healthy side of the PFPS group (40 knees) and both side of the healthy control group (80 knees). Randomization was applied with random-number generator (Research Randomizer. Version 4.0). Only one of the authors was aware of randomization. Examiner and patient were blind to the relevant group. Non-selective closed kinetic chain and selective closed kinetic chain exercises were applied for 6 weeks in all groups. Thigh circumference measurement was performed 5-10 cm above the upper pole of the patella. In addition, evaluation was made with visual analog score (VAS) and Lysholm Knee Score (LKS) score. Vastus medialis obliquus (VMO) and vastus lateralis (VL) muscles of the participants were measured with Shear Wave Elastography 1 day before the therapy and 6 weeks after therapy. Written informed consent was taken from each patient.This study is in line with the Declaration of Helsinki. Approval was obtained by the Local Ethics Committee (17/07/2016-258642).

ELIGIBILITY:
Inclusion Criteria:

* Having peripatellar/retropatellar pain while sitting,going up and down the stairs
* Walking for a long time, crouching down, running, and kneeling down
* Having a VAS score of ≥3 during the evaluation and not developing these symptoms on a traumatic basis

Exclusion Criteria:

* Tendinitis
* Osgood-Schlatter Syndrome
* Traumatic hip or knee injuries
* Osteoarthritis
* Plica syndrome
* Sinding-Larsen-Johansson syndrome
* Ligamentous instability
* Spinal pain
* Chondral lesion
* Patellar tendon pathology
* Distraction apophysitis of knee circumference

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Shear Wave Elastography | 1 day before exercise program
  Measurement of muscle strength before exercises
Shear Wave Elastography | 6 weeks after exercise program
  Measurement of muscle strength after exercises

REFERENCES:
- [Derived] Kultur Y, Harbiyeli E, Botanlioglu H, Ozsahin MK, Ozturhalli S, Aydingoz O, Erginer MR. Evaluation of the results of closed kinetic chain exercises applied in the conservative treatment of patellofemoral pain syndrome by means of shear wave elastography: A randomized controlled trial. J Orthop Surg (Hong Kong). 2024 Sep-Dec;32(3):10225536241280384. doi: 10.1177/10225536241280384. PMID 39483049